CLINICAL TRIAL: NCT05769049
Title: A Randomized, Observer-Blinded, Active-Controlled, Phase I Study to Evaluate the Safety and Immunogenicity of the Recombinant Zoster Vaccine (CHO Cell) in Healthy Adults Aged 40 Years and Older
Brief Title: The Safety and Immunogenicity Study of the Recombinant Zoster Vaccine (CHO Cell)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Rec-Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REC610C102
Record Dates: First submitted 2023-01-27; First posted 2023-03-15 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Intervention Model Description: Totally 48 eligible participants, 24 for each age group, will be enrolled in the study with a 2:1 randomization ratio to receive REC610 (50 μg) or Shingrix® (50 μg) respectively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REC610 (Experimental): Lyophilized gE antigen: white cake or powder. clear to opalescent, colorless liquid after reconstitution with water for injection BFA01 adjuvant suspension: opalescent white liquid After reconstitution: opalescent white liquid. Each dose (0.5 mL) contains 50 μg of Quillaja Saponin (QS-21), 50 μg of MPL, 1 mg of dioleoyl phosphatidylcholine, and 0.25 mg of cholesterol
  Interventions: Biological: REC610
- Shingrix (Active Comparator): Lyophilized gE antigen: white cake or powder. clear to opalescent, colorless liquid after reconstitution with water for injection AS01B adjuvant suspension: opalescent, colorless to pale brownish liquid suspension After reconstitution: opalescent, colorless to pale brownish liquid. Each dose (0.5 mL) contains 50 μg of QS-21, 50 μg of MPL, 1 mg of dioleoyl phosphatidylcholine, and 0.25 mg of cholesterol
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: REC610 — administered as 2 intramuscular (IM) injections in healthy adults aged 40 years and older
  Other Names: Recombinant Zoster Vaccine (CHO cell)
  Arms: REC610
Biological: Shingrix — Shingrix
  Other Names: Recombinant Zoster Vaccine (CHO cell)
  Arms: Shingrix

SUMMARY:
This is a randomized, observer-blinded, active-controlled Phase I study to evaluate the safety, reactogenicity, and immunogenicity of REC610, when administered as 2 intramuscular (IM) injections in healthy adults aged 40 years and older, who do not have known HZ and history of varicella or HZ vaccination. The recombinant HZ vaccine, Shingrix® (GlaxoSmithKline), will be used as the active control.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and reactogenicity of REC610, and the secondary objective is to evaluate the immunogenicity of REC610.

The study will include younger (40 to 59 years, included) and older (60 years and above) healthy adult participants in 2 separate age groups. Totally 48 eligible participants, 24 for each age group, will be enrolled in the study with a 2:1 randomization ratio to receive REC610 (50 μg) or Shingrix® (50 μg) respectively. The study will progress in a sequential manner, with the younger adult group being enrolled and vaccinated first.

The Safety Monitoring Committee (SMC) will review the safety data after all participants in the younger adult group complete the 7 days visit after the first vaccination. The older adult enrollment will commence only after the SMC's review is completed.

Participants will undertake a Screening Visit between Day -7 and Day -1 to determine their eligibility. The eligible participants will be randomized to receive the first dose vaccination on Day 0, and the second dose vaccination at 60 days (+14 days) post the first dosing, according to the allocated group. Verification on the criteria for vaccination postponement or termination should be performed before the second dosing. Additionally, all the participants will return to the study site for ongoing assessments of safety and immunogenicity as per the Schedule of Assessments Visits.

Sentinels will be employed for each age group during the first dose vaccination. Each age group will include 3 sentinel participants (2 REC610, 1 Shingrix®) who will be dosed first and monitored by the Investigator for at least 2 hours at the study site; discharge will only be allowed per agreement by the Investigator. After 48 hours post the study vaccination, the sentinel participants will be contacted by site staff via telephone/text message/other mode to collect and record AEs. Once the dose is deemed to be safe by the absence of significant safety issues in the sentinels, in consultation with the study Medical Monitor and Sponsor as needed, the remaining participants in the age group will be randomized (2:1) to receive REC610 or Shingrix®, respectively. The decision to dose the rest of the age group will be documented.

All participants will be followed up for safety and reactogenicity. Participants will be observed for 30 minutes at study site after each dosing. For the sentinels, the observation requires to be at least 2 hours post the first dosing. Before leaving the study site, participants will be given diaries and be trained on recording solicited AEs within 7 days and unsolicited AEs within 30 days after each dosing. All participants will return to study site on Day 7 (+3 days) for safety clinical laboratory assessment. Besides, the occurrence of SAEs and AESIs will be monitored from the first dose vaccination till 6 months after the second dose vaccination.

In addition, all participants will be followed up for immunogenicity. Blood samples will be collected on Day 0 (before the study vaccination), at 60 days after the first dose vaccination (+14 days, before the second dose vaccination), 30 days (+7 days), 3 months (+15 days), and 6 months (+30 days) after the second dose vaccination, respectively, for testing of gE specific antibodies and assessing on the cellular immune response. Blood samples will be sent to the central laboratory for the immunogenicity testing.

During the whole study period, if participants have any signs or symptoms related to HZ, the diagnosis and necessary management will be performed per local clinical practice at the study site. After HZ diagnosis is confirmed, the participants will receive safety follow-up only during the leftover study stage.

Interim Analysis & Final Analysis The interim analysis (IA) is planned after all participants complete 30 days visit post the second dose vaccination, to evaluate safety and immunogenicity during this period. The IA for each age group may be conducted separately, depending on the actual enrollment progress. The IA will be performed by an independent statistic group, while the sponsor will be kept blinded from participant's individual randomization information. The investigators, all study participants and study team members except for unblinded staff assigned for IPs management and monitoring at site, will be kept blinded during the entire study period. The results of IA will support the design on following clinical trials for REC610. Within the IA, all the study procedures for long-term follow-up will be continued.

The Final Analysis (FA) will be conducted after all participants complete the follow-up visit at 6 months after the second dose vaccination, to evaluate long-term safety and immune persistency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40 years and older.
* Able and willing to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteers' medical history with his/her general practitioner/personal doctors and access all medical records which are relevant to study procedures.
* Healthy adults, or adults with stable medical condition who have a pre-existing medical condition that does not meet any exclusion criteria. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.

Exclusion Criteria:

* Known history of COVID-19 within 6 months prior to randomization, or being defined as SARS-CoV-2 infection by RT-PCR assay during the screening.
* Fever (oral temperature ≥ 37.5°C / axillary temperature ≥ 37.3°C) on the day of vaccination, or having fever within recent 72 hours before the vaccination.
* Known history of herpes zoster.
* History of varicella or herpes zoster vaccination.
* Having abnormal results of clinical laboratory testing during screening, which is judged by the investigator with clinical significance, including the hematology, blood chemistry, and urinalysis.
* History of severe allergic diseases or reactions likely to be exacerbated by any component of investigational vaccine, including the adjuvant components (e.g., QS-21, MPL, common in foamer for beverage, emulsive flavor composition, vitamin E, mildew preventive, and part of Chinese herbal medicine, e.g., ginseng, balloon-flower root, liquorice), such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local hypersensitive necrosis reaction (Arthus reaction), prior history of serious adverse reaction to any vaccine or drug, such as acute allergy, urticaria eczema, dyspnea, and angioneurotic edema.
* Having malignant tumors (except for skin basal cell carcinoma or carcinoma uterine cervix in situ), immune diseases (e.g., known documented human immunodeficiency virus [HIV] infection, systemic lupus erythematosus, rheumatoid arthritis, alienia or splenectomy, and others that may influence immune response at the investigator's discretion).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Incidence of related AE | within 30 days after each dose vaccination
  The incidence of investigational product (IP)-related adverse events (AEs) within 30 days after each dose vaccination.
Incidence of solicited AE | within 7 days after each dose vaccination
  The incidence of solicited local and systemic AEs within 7 days after each dose vaccination.
Incidence of unsolicited AEs | within 30 days after each dose vaccination
  The incidence of unsolicited AEs within 30 days after each dose vaccination.
Incidence of clinically significant abnormalities in clinical laboratory tests | Day 7 after the first dose vaccination
  The incidence of clinically significant abnormalities in clinical laboratory tests (hematology, blood chemistry, and urinalysis) on Day 7 after the first dose vaccination
Occurrence of serious adverse events (SAEs) and adverse events of special interests (AESIs) | 6 months after the second dose vaccination
  The occurrence of serious adverse events (SAEs) and adverse events of special interests (AESIs) till 6 months after the second dose vaccination

SECONDARY OUTCOMES:
The seroconversion rate (SCR) at timepoints during the study | 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination
  The seroconversion rate (SCR) of glycoprotein E (gE) specific antibody at 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination.
The geometric mean titer (GMT) at timepoints during the study | 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination
  The geometric mean titer (GMT) of glycoprotein E (gE) specific antibody at 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination.
The geometric mean increase (GMI) at timepoints during the study | 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination
  The geometric mean increase (GMI) of glycoprotein E (gE) specific antibody at 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination.
Frequencies of CD4+ T cells secreting at least one of gE specific cytokines (e.g., IFN-γ, IL-2, TNF-α, CD40L) per 106 CD4+ T cells, and the cell mediated immunity (CMI) response rates at timepoints during the study | 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination
  The frequencies of CD4+ T cells secreting at least one of gE specific cytokines (e.g., IFN-γ, IL-2, TNF-α) per 106 CD4+ T cells, and the cell mediated immunity (CMI) response rates at 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination.
Frequencies of CD4+ T cells secreting at least two of gE specific cytokines (e.g., IFN-γ, IL-2, TNF-α) per 106 CD4+ T cells, and the cell mediated immunity (CMI) response rates at timepoints during the study | 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination
  The frequencies of CD4+ T cells secreting at least two of gE specific cytokines (e.g., IFN-γ, IL-2, TNF-α, CD40L) per 106 CD4+ T cells, and the cell mediated immunity (CMI) response rates at 60 days after the first dose vaccination (before the second dose vaccination), 30 days, 3 months and 6 months after the second dose vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Loreta Zoleta- De Jesus, Dr., Principal Investigator — Silang Specialists Medical Center
Locations (1):
- Pharma Peak Research Philippines,Inc., Makati City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.